CLINICAL TRIAL: NCT05935592
Title: Intervention INC: An Interactive Family-centered mHealth Tool to Reduce Obesity Risk in Urban Minority Preadolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Children's Aid, New York City (Unknown); Washington University School of Medicine (Other); Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency); Hunter College of City University of New York (Other); City University of New York, School of Public Health (Other); University of Massachusetts, Amherst (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00004065; 5R01HS028650-03 (AHRQ)
Record Dates: First submitted 2023-06-29; First posted 2023-07-07 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2024-10

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): The experimental group will receive access to Intervention INC, a theory-guided interactive, family-centered web-based tool promoting healthy dietary behaviors.
  Interventions: Behavioral: Web-based comic and newsletters
- Comparison Group (Active Comparator): The comparison group will receive access to web-based newsletters focused on promoting healthy dietary behaviors.
  Interventions: Behavioral: Didactic health information

INTERVENTIONS:
Behavioral: Web-based comic and newsletters — Web-based comic and health messages (child component) and health newsletters (parent component)
  Arms: Experimental Group
Behavioral: Didactic health information — Web-based newsletters (for child and parent) by email and/or text
  Arms: Comparison Group

SUMMARY:
Using a two-group randomized study design, this study aims to evaluate the effectiveness of the adapted family-centered mHealth tool on child BMI z-score (primary outcome), child dietary behaviors, and parental feeding practices, from baseline to 12-month follow-up, among 200 child-parent dyads. It is hypothesized that children in the experimental group will demonstrate larger BMI-z score improvements between baseline and 12-month follow-up compared to children in the comparison group.

DETAILED DESCRIPTION:
Childhood obesity continues to be a serious clinical and public health issue in the United States (US), particularly within low-income, minority groups. Effective, yet engaging interventions, such as the one developed by our team, are needed to capture the attention of children living in a multi-media environment.

Potentially eligible pediatric patients (and their parent/caregiver) will be recruited from two of Children's Aid community-based clinics in NYC - Dunlevy Milbank Center based in Harlem and the Bronx Health Center based in the South Bronx. A variety of recruitment methods will be deployed, including in-person/flyer-based recruitment in clinic waiting rooms, healthcare provider referrals, and direct calls.

At baseline, eligible participants will be randomized to either the experimental group or comparison group (allocation ratio 1:1). Randomization will be performed at the dyad level and will be balanced on child ethnicity (Hispanic or Non-Hispanic), child biological sex (male, female), and clinic site.

The experimental group will receive access to Intervention INC, a theory-guided interactive, family-centered web-based tool promoting healthy dietary behaviors. The comparison group will receive access to web-based newsletters focused on promoting healthy dietary behaviors. To minimize bias, participants will be blinded to the study's hypothesis.

Data will be collected at four timepoints: baseline (T1), main intervention end (T2), maintenance intervention end (T3), and at 12-month follow-up (T4). The primary outcome measure (BMI z-score) will be calculated using height and weight data captured via combined scale/stadiometer by a trained healthcare provider at T1, T3, T4. Secondary measures (dietary intake and dietary knowledge & attitudes of child participants; feeding practices and the home food environment by the parent/caregiver) will be captured via questionnaires at T1, T2, T3, T4.

ELIGIBILITY:
Inclusion Criteria (child):

* self-identifies as Black/African-American and/or Latino
* between ages 8 and 12 years (preadolescents) at time of scheduled baseline visits
* reads and speaks in English
* has a Body Mass Index percentile at or above 5% at baseline (categorized as healthy, overweight, or obese)
* has regular internet access via a tablet device, smartphone, or computer/laptop
* has regular access to a phone with texting capability
* is comfortable reading/viewing material on electronic devices
* is comfortable speaking with study staff about thoughts/experiences while participating in study
* has a legal parent/guardian willing to participate in study

Inclusion Criteria (parent):

* legal parent/guardian of child willing to participate in study
* reads and speaks in English or Spanish
* primarily responsible for preparing/purchasing food for child
* has regular internet access via a tablet device, smartphone, or computer/laptop
* has regular access to a phone with texting capability
* comfortable reading/viewing material on electronic devices
* able to attend in-person study visits and complete online questionnaires with their child over the full duration of study

Exclusion Criteria (child):

* has allergies, food aversions, food disorders, or medications with side-effects that may impact participation in study
* has a pacemaker or heart condition
* in foster care

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in BMI z-score | T1 (baseline), T3 (maintenance intervention end, 6 months post-T2), T4 (follow-up, 12 months post T2)
  BMI z-score calculation based on measured height and weight

SECONDARY OUTCOMES:
Change in child dietary intake | T1 (baseline), T2 (intervention end, 12-weeks post-baseline), T3 (maintenance intervention end, 6 months post-T2), T4 (follow-up, 12 months post T2)
  17-item questionnaire completed by child participants assessing frequency of consumption of fruit/vegetables, water, junk food, and sugary drinks during the past seven days
Change in child dietary knowledge and attitudes | T1 (baseline), T2 (intervention end, 12-weeks post-baseline), T3 (maintenance intervention end, 6 months post-T2), T4 (follow-up, 12 months post T2)
  45-item questionnaire completed by child participants assessing knowledge, outcome expectations, self-efficacy, and behavioral intention regarding behaviors associated with fruit/vegetables, water, junk food, and sugary drinks
Change in parent feeding practices | T1 (baseline), T2 (intervention end, 12-weeks post-baseline), T3 (maintenance intervention end, 6 months post-T2), T4 (follow-up, 12 months post T2)
  27-item questionnaire completed by parent participants assessing multiple parental feeding practices
Change in home food environment | T1 (baseline), T2 (intervention end, 12-weeks post-baseline), T3 (maintenance intervention end, 6 months post-T2), T4 (follow-up, 12 months post T2)
  6-item questionnaire completed by parent participants assessing availability of fruits/vegetables and water in their home and how often they store fruits/vegetables and water in a place easily seen by their child

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Milbank Health Center - Children's Aid, New York, New York
  - Bronx Health Center - Children's Aid, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No